CLINICAL TRIAL: NCT06941519
Title: Addressing Social Needs to Improve Health in Adults With Multiple Chronic Conditions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: IRB 2291224; BPS-2023C3-35937 (Other Grant/Funding Number: Patient Centered Outcomes Research Institute)
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-04

CONDITIONS: Multiple Chronic Conditions; Social Needs; Care Gaps; Navigation
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telephonic Navigation (Experimental): Higher Intensity (active telephonic outreach from a health navigator with follow-up contacts for up to 3 months)
  Interventions: Behavioral: Telephonic Outreach
- Virtual Outreach (Active Comparator): Lower Intensity (outreach via text, email, and/or letter with materials that contain information about available local, state, and federal governmental benefits and services)
  Interventions: Behavioral: Virtual Outreach

INTERVENTIONS:
Behavioral: Telephonic Outreach — Higher Intensity (active telephonic outreach from a health navigator with follow-up contacts for up to 3 months)
  Arms: Telephonic Navigation
Behavioral: Virtual Outreach — Lower Intensity (outreach via text, email, and/or letter with materials that contain information about available local, state, and federal governmental benefits and services)
  Arms: Virtual Outreach

SUMMARY:
The investigators will conduct a comparative effectiveness randomized clinical trial with two "active comparator" arms. The investigators will evaluate the two current, usual care strategies (higher intensity "telephonic navigation" vs. lower intensity "virtual outreach") for addressing social needs among patients with multiple chronic conditions.

DETAILED DESCRIPTION:
The goal of the proposed research is to compare the effectiveness of two strategies for addressing social needs in a large, high-risk population of adults with multiple chronic conditions (MCC).

Specific Aims are to:

Aim 1 - Comparative Effectiveness Randomized Clinical Trial: Compare two evidence-based strategies for systematically addressing patient-reported social needs in a medically complex population: Higher Intensity (active telephonic outreach from a health navigator with follow-up contacts for up to 3 months) vs. Lower Intensity (outreach via text, email, and/or letter with materials that contain information about available local, state, and federal governmental benefits and services). Hypotheses (H) are framed in terms of relatively greater effectiveness of the Higher Intensity strategy, although through Aims 2 & 3 the investigators will investigate variation within different patient groups.

H1: Overall improvement will be greater in the Higher vs Lower Intensity strategy condition on the primary (receipt of social services, social needs met, clinical care gaps closed) and secondary (patient-centered) outcomes.

Aim 2 - Qualitative Assessment: The investigators will conduct patient focus groups and navigator interviews to examine intervention impact and mechanisms at each step in the pathway from intervention engagement to obtaining social resources to addressing social needs to improving clinical care and to explore associated barriers and facilitators. Exploratory Qualitative Hypotheses (QH) are:

QH1: Patients will describe greater perceived impacts and positive experiences in the high intensity intervention condition than the low intensity intervention condition.

QH2: Patients and navigators will describe both direct pathways by which social risk screening and/or receipt of referrals impacts chronic disease (e.g., improved social resources) as well as indirect pathways (e.g., reduced stress, fewer competing demands, improved trust due to patient-provider/navigator relationship, increased medication affordability and use.)

Aim 3 - Heterogeneity of Treatment Effects (HTE): The investigators will test the hypothesis that one or other of the two interventions is more impactful within prespecified sub-groups based on patient factors (age, type of social need, educational attainment) and clinical factors (comorbidity, care gaps) to inform strategies for future adaptation and dissemination.

HTE hypotheses: Younger age, higher educational attainment, fewer social needs, fewer chronic conditions, fewer care gaps will each be associated with better outcomes in the Lower Intensity vs Higher Intensity intervention arms.

Cumulatively, these three aims will provide timely and policy-relevant comparative effectiveness evidence to inform health care system approaches to addressing social needs in patients with chronic conditions (Aim 1), to understand mechanisms of action and key design elements from patient and navigator perspectives along the pathway from screening to improved health (Aim 2), and to investigate differential impacts across sub-populations (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

* Two or more chronic medical conditions from a defined list of 24 chronic conditions
* One or more gaps in evidence-based care (related to condition-specific risk factor management, evidence-based screening and preventive care, missed appointments, and medication non-adherence),
* At least one self-reported social-related barrier to care or "social need" (e.g., transportation, food, housing, utilities, and/or financial insecurity).

Exclusion Criteria:

* major cognitive barriers (dementia, psychosis).
* multiple prior year hospitalizations ("extremely high utilizers")

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2029-09-15 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Receipt of social services | approximately 6 months after enrollment
  Patient survey re: receipt of resources from available programs
Reduction in number of social needs | approximately 6 months after enrollment
  Reduction from baseline in number of unmet social needs
Clinical care gap closure | approximately 12 months after enrollment
  Reduction in number of evidence-based clinical care gaps

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Grant, MD MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- Division of Research, Pleasanton, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tucher EL, Steele AL, Uratsu CS, Hamilton LK, Brown MC, Nugent JR, Jones DH, Gottlieb LM, Grant RW. Addressing social needs to improve health in adults with multiple chronic conditions: A comparative effectiveness trial of two real-world social needs interventions. Contemp Clin Trials. 2025 Dec 24;161:108210. doi: 10.1016/j.cct.2025.108210. Online ahead of print. PMID 41453516